CLINICAL TRIAL: NCT06731855
Title: An Exploratory Physiological Study of Post-operative Recovery in Surgical Neonates and Dimethylarginine:Arginine Levels (SuNDiAL)
Brief Title: An Exploratory Physiological Study of Post-operative Recovery in Surgical Neonates and Dimethylarginine:Arginine Levels
Acronym: SuNDiAL
Status: Recruiting | Type: Observational
Sponsor: Liverpool Women's NHS Foundation Trust (Other)
Collaborators: Alder Hey Children's NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 349681
Record Dates: First submitted 2024-12-09; First posted 2024-12-12 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2024-12

CONDITIONS: Gastroschisis; Congenital Diaphragmatic Hernia; Duodenal Atresia; Oesophageal Atresia With Tracheo-Oesophageal Fistula; Oesophageal Atresia; Exomphalos
Keywords: Neonatal; Abdominal Surgery; Asymmetric Dimethylarginine; ADMA; Arginine; Recovery; Neonate
MeSH Terms: conditions — Gastroschisis; Hernias, Diaphragmatic, Congenital; Familial duodenal atresia; Esophageal atresia with or without tracheoesophageal fistula; Esophageal Atresia; Hernia, Umbilical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Study Population: Infants born >35 weeks gestation and have a condition requiring major gastrointestinal surgery within 5 days (120 hours) of birth. This is expected to include predominantly congenital gut malformations such as gastroschisis, gut atresias, volvulus and congenital diaphragmatic hernia (who are stable enough for surgery in this time frame).
  Interventions: Procedure: Abdominal Surgery for congenital gut malformation in the first 5 days of life.

INTERVENTIONS:
Procedure: Abdominal Surgery for congenital gut malformation in the first 5 days of life. — Abdominal Surgery for congenital gut malformation in the first 5 days of life. Procedure will depend on the congenital gut malformation.

SUMMARY:
The SuNDiAL study will measure levels of two naturally occurring amino acids: Arginine and Asymmetric Dimethylarginine (ADMA) in neonates undergoing abdominal surgery in the first 5 days of life due to congenital abdominal malformations as the participants recover from surgery.

The investigators hypothesise that the relationship between Arginine and ADMA may be useful in predicting recovery and complications in babies who have had abdominal surgery due to previous research published in adult patients undergoing abdominal surgery. If this relationship is found to be useful there may be options for developing treatments (such as arginine supplementation) in the future to improve recovery and reduce complications in neonates undergoing abdominal surgery.

Neonates born after 35 weeks gestation who have a congenital abdominal malformation who require abdominal surgery in the first 5 days will be eligible to participate in the SuNDiAL study.

Arginine and ADMA will be measured from blood samples that are left over from the participant's blood tests that are taken as part of their routine clinical care. The investigators will measure Arginine and ADMA preoperatively and at least 10 points in the 30 days following their surgery, or until the participant fully recovers from surgery (which ever comes first). There is no intervention in the SuNDiAL study, and there will be no extra blood or blood samples taken.

Serums samples that are left over from the babies routine clinical blood tests will be stored securely in the hospitals laboratory until analysis for Arginine and ADMA.

The levels of Arginine and ADMA will be compared to the time it takes the participants to recover from surgery and any complications that may arise following surgery. During the study the study team will use the participants electronic medical record to establish when the participant became fully established on oral feeding and monitor for any complications that occurred during their recovery.

DETAILED DESCRIPTION:
The study is a prospective observational, physiological study running across the two trust that form the Liverpool Neonatal Partnership; Liverpool Women's Hospital NHS Foundation Trust and Alder Hey Children's Hospital Foundation Trust.

There is no study intervention and therefore all participants will be managed in accordance with existing local protocols and current accepted clinical practice. Participants will receive standard neonatal and surgical care as per the local clinical guidelines. The participant will have routine blood tests taken as part of their routine care. No additional blood or blood tests will be taken for the SuNDiAL study.

The study will involve the analysis of any blood left over from samples taken routinely pre and postoperatively in infants who have undergone abdominal surgery. Residual serum samples will be analysed from the blood samples taken for routine blood monitoring in the infants enrolled in the study. Biochemical samples will undergo Enzyme-linked immunosorbent assay (ELISA) analysis for ADMA and arginine.

The study period is from preoperatively until 30 days post operatively or until the baby fully recovers from surgery, marked by being fully fed with milk into their stomach. The aim is to obtain at least 1 measurement preoperatively, and a minimum of 4 measurements in the post-operative period. The expectation is that 3-5 measurements first 10 postoperative days should be achievable.

The SuNDiAL study will aim to determine if the level of ADMA and/or Arginine and/or the Arginine to ADMA ratio is associated with the time taken to recover following major abdominal surgery in neonates born after 35 weeks gestation. Recovery will be measured as the time taken to no longer require intravenous nutrition following surgery as the primary objective.

The secondary objectives include:

1. To develop a mathematical model of postoperative ADMA and/or ARG/ADMA ratio. This will allow future randomised controlled trial designs investigating postoperative recovery time to include ADMA and ARG/ADMA in the study protocol. This modelling has the potential to develop future arginine supplementation protocols to target and/or refine arginine dosage and duration based on the trajectory of the ADMA levels or arginine:ADMA ratio. This approach includes specific post operative complications following surgery that may delay recovery (such as mortality, wound healing, sepsis, parenteral nutrition cholestasis)
2. To compare ADMA and/or ARG/ADMA ratio in specific gastrointestinal conditions that require major abdominal surgery.
3. To assess ADMA and the ARG/ADMA ratio in specific gastrointestinal conditions that require major abdominal surgery, pre and postoperatively.
4. To identify whether amino acid (protein) and/or arginine intake affect plasma ADMA levels in the post-operative period and to incorporate this outcome in future randomised controlled trials investigation arginine supplementation and other nutritional interventions.

Parents of potential participants will be approached preoperatively or up to 5 days postoperatively to complete the informed consent process.

Once the parents of potential participants have had sufficient time to read and process the information regarding the study (minimum 2 hours), and sufficient time to ask questions regarding the study, written consent will be obtained.

Blood samples will be taken by the clinical team routinely as part of their clinical care. Patients will be managed as per accepted clinical practice and local clinical guidelines by the clinical team. There will be no changes from routine practice due to the SuNDiAL study. No extra blood tests will be taken for the SuNDiAL study.

If an infant is eligible and the parents have given consent to participate in the SuNDiAL study, at the time of ordering routine clinical blood tests the clinical team will order an additional dummy blood test 'SUNDIAL store sample'.

If there is any remaining serum following routine clinical blood tests, the 'SUNDIAL store sample' will alert the lab to store the blood sample for the SuNDiAL study. The sample will frozen and be stored in the SuNDiAL area of the research laboratory freezer in Alder Hey Children's Hospital. All samples with serum remaining will be stored. Samples will stop being stored once the patient is fully recovered or after 30 days post operatively which ever occurs first. The sample will be available for the clinical team to do further tests if these are required and this will take priority over testing the blood for research purposes.

Once there is sufficient samples to run an analysis the samples with be transported to the research laboratory. The samples will then be analysed by the ELISA technique, to measure Arginine and ADMA. Samples will be anonymised by the research team prior to being transported to the Research Laboratory in the Institute in the park at Alder Hey Children hospital.

The data will be anonymised prior to analysis. Data will be analysed for both the primary and secondary outcomes outlined above by the University of Liverpool Computational Biological Facility.

ELIGIBILITY:
Inclusion Criteria:

1. Infants born >35 weeks gestation
2. Have a condition requiring major gastrointestinal surgery
3. Surgery within the first 5 days (120 hours) following birth (including congenital diaphragmatic hernia who are stable enough for surgery in this time frame).
4. Parent(s)/guardian(s) must have a comprehensive understanding of written and spoken English, sufficient to provide informed using the translation services available to the research team.
5. Must be willing and able to provide informed consent in order to take part in the study

Exclusion Criteria:

1. Infants who are unlikely to survive because of poor immediate postoperative condition.
2. Infants known (or suspected to have) a diagnosis of inborn error of metabolism or serious liver dysfunction.
3. Parent(s)/guardian(s) who are unable to give informed consent.
4. Infants who it is not possible to obtain the minimum required residual serum samples from routine biochemical blood testing as outlined in the study schedule

Max Age: 5 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population with be of 30 infants born >35 weeks gestation and has a condition requiring major gastrointestinal surgery within 5 days (120 hours) of birth. This is expected to include predominantly congenital gut malformations: gastroschisis, gut atresias, volvulus and congenital diaphragmatic hernia (who are stable enough for surgery in this time frame).
  Patient will be recruited over a 1 year period. These infants will be born at Liverpool Women's Hospital or at their local hospital in the north west of England region, and transferred to Alder Hey Children's Hospital for their operation, either directly or via Liverpool Women's Hospital Neonatal Intensive Care Unit. They will recover in Alder Hey Children's Hospital's Paediatric Intensive Care Unit or Neonatal Surgical Unit and may later be transferred back to Liverpool Women's Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-02-05 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
The relationship between Arginine, ADMA and the Arginine to ADMA ratio in comparison to the time taken to recover from abdominal surgery. | From Enrolment to 30 days following surgery
  The primary outcome measure will investigate the level of plasma ADMA, arginine and ARG/ADMA ratio preoperatively and in the immediate postoperative period (5 days) in infants stratified according to typical (<21 days) or prolonged (>21 days) postoperative PN dependency. The following measures will be compared between the typical and prolonged recover groups:
  1. The pre-operative level (peak/trough as appropriate) of Arginine, ADMA and the ARG/ADMA ratio.
  2. The post-operative level (peak/trough as appropriate) within 5 days of surgery of arginine, ADMA and the ARG/ADMA ratio and its relationship to postoperative PN days.
  3. The maximum per-infant difference between pre-operative and post-operative levels as defined in a) and b).

SECONDARY OUTCOMES:
Develop a mathematical model to describe the entire postoperative (30 days) trajectory of Arginine, ADMA and the ARG/ADMA ratio in relation to PN dependency. | From enrolment until day 30 post operatively.
To study the relationship over time between nutritional intake and arginine, ADMA and the ARG/ADMA ratio. | From enrolment until day 30 postoperatively.
The relationship over time between clinically monitored postoperative inflammatory and biochemical markers and arginine, ADMA and the ARG/ADMA ratio | From Enrolment to 30 days post operatively
Impact of individual episodes (including duration) of any recognised postoperative complication (eg wound complications, bowel complications, sepsis) on the recovery time and the mathematical model described above. | From enrolment to 30 days post operation
Weight Gain/head growth over the study period in relationship to Arginine, ADMA and Arginine to ADMA ratio. | Enrolment to 30 days post operation.
Level of care and major treatments (eg ventilation, inotropic support, antibiotics for sepsis) during the study period in relation to Arginine, ADMA and the Arginine to ADMA ratio. | From enrolment to 30 days postoperatively.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Alder Hey Childrens Hospital NSH Foundation Trust, Liverpool, Merseyside
  - Liverpool Womens Hospital NHS Foundation Trust, Liverpool, Merseyside

IPD SHARING:
Plan to Share IPD: No